CLINICAL TRIAL: NCT00510588
Title: Chronic Inflammatory Activation in Fat Tissue: an Atherogenic Factor in Stable Coronary Artery Disease
Acronym: KFO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Robert Hoellriegel, Co-Investigator, University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0815-2007
Record Dates: First submitted 2007-08-01; First posted 2007-08-02 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Stable Coronary Artery Disease; Obesity; Impaired Glucose Tolerance
Keywords: adiposity
MeSH Terms: conditions — Obesity; Glucose Intolerance | interventions — Metformin

ARMS (4):
- 1 (Other): regular physical exercise training
  Interventions: Other: training
- 2 (Other): regular physical exercise training + metformin
  Interventions: Other: training + metformin
- 3 (Other): regular physical exercise training + glitazon
  Interventions: Other: training + glitazon
- 4 (No Intervention): Control

INTERVENTIONS:
Other: training — regular physical exercise training for 6 months
  Arms: 1
Other: training + metformin — regular physical exercise training in combination with metformin for 6 months
  Arms: 2
Other: training + glitazon — regular physical exercise training in combination with a glitazon for 6 months
  Arms: 3

SUMMARY:
Chronic inflammatory activation in fat tissue can be the link between adiposity and an increased risk for atherosclerosis. Aim of the study is to investigate how molecular alterations in fat tissue can be influenced by regular physical exercise training alone or in combination with a medical therapy (Glitazon or Metformin) in obese patients with stable CAD and impaired glucose tolerance.

ELIGIBILITY:
Inclusion Criteria:

* either impaired glucose tolerance (2-h plasma glucose concentration >7.8 and <11.1 mmol/L during an oral glucose tolerance test) or impaired fasting glucose (fasting glucose concentration >6.0 and <7.0 mmol/L)
* coronary artery disease determined by coronary angiography
* BMI > 25
* male patients aged 35-75 years

Exclusion Criteria:

* diabetes mellitus type 1
* diabetes mellitus type 2 in combination with glycosylates hemoglobin >6.0%, previous medication with oral antidiabetic agents or insulin, fasting plasma glucose concentration > 11.0 mmol/L
* unstable angina pectoris
* indication for coronary artery bypass graft operation
* myocardial infarction within the last 3 months
* reduced left-ventricular systolic function < 40 %

Ages: 35 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2007-07; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
change in endothelial function in patients with stable coronary artery disease | 6 months

SECONDARY OUTCOMES:
change in metabolic parameters | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Schuler, Prof. of medicine, Principal Investigator — Heart Center Leipzig - University Hospital
Locations (1):
- University of Leipzig - heart center, Leipzig, Germany